CLINICAL TRIAL: NCT04583046
Title: Effects of Iloprost on Pulmonary Oxygenation in Obese Patients During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2020-0722
Record Dates: First submitted 2020-09-17; First posted 2020-10-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Including Metastatic Cancer); Pulmonary Infection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): normal saline inhalation group
  Interventions: Drug: normal saline inhalation
- iloprost group (Experimental): iloprost inhalation group
  Interventions: Drug: iloprost inhalation

INTERVENTIONS:
Drug: normal saline inhalation — When anesthesia induction finishes, change patients' position from supine to lateral position and measure ABGA, VBGA while two lung is ventilated (T0). After 20 minutes of applying one-lung ventilation, measure ABGA and VBGA (T1). Apply normal saline inhalation for control group and measure ABGA at the time of 20 min after normal saline inhalation has finished (T2).
  Arms: placebo
Drug: iloprost inhalation — When anesthesia induction finishes, change patients' position from supine to lateral position and measure ABGA, VBGA while two lung is ventilated (T0). After 20 minutes of applying one-lung ventilation, measure ABGA and VBGA (T1). Apply iloprost inhalation for iloprost group and measure ABGA at the time of 20 min after iloprost inhalation has finished (T2).
  Arms: iloprost group

SUMMARY:
One lung ventilation (OLV) is essential during thoracic surgery. During OLV, intrapulmonary shunt can be increased resulting hypoxemia. Although OLV technique had been advanced so far, hypoxemia during OLV reaches about 10% in spite of inspired oxygen fraction 100%. Iloprost is a prostaglandin analogue used for pulmonary hypertension, which can decrease pulmonary artery resistance by selectively dilating pulmonary artery. In this prospective, randomized, double blind study, the investigator is planning to investigate the effects of iloprost on respiratory physiology (intrapulmonary shunt, deadspace, oxygenation, etc) in obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. scheduled for VATS lobectomy
2. 40 < age < 80
3. American Society of Anaesthesiologists(ASA) physical status classification I~III
4. BMI > 30 kg /m2

Exclusion Criteria:

1. American Society of Anaesthesiologists(ASA) physical status classification IV or more
2. NYHA class III~IV
3. Severe obstructive lung disease and/or restrictive lung disease patients
4. patients with end-organ diseases (i.e. heart failure, respiratory failure, hepatic failure, renal failure)
5. arrhythmia
6. pregnant women
7. pulmonary edema or pulmonary arterial hypertension
8. cerebrovascular disease
9. unstable angina or myocardial infarction within 6 months
10. patients with allergic reaction at iloprost

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Result of arterial blood gas analysis : partial pressure of oxygen(PaO2) | 20 minutes after iloprost inhalation (T2)
Result of arterial blood gas analysis : partial pressure of oxygen in the arterial blood(PaO2)/Fraction of inspired oxygen(FiO2) ratio (P/F ratio) | 20 minutes after iloprost inhalation (T2)
Result of arterial blood gas analysis : Oxygen saturation in arterial blood(SaO2) | 20 minutes after iloprost inhalation (T2)

SECONDARY OUTCOMES:
deadspace | 20 minutes after iloprost inhalation (T2)
  Dead space ventilation was calculated with Paco2 and end-tidal carbon dioxide (Etco2) according to the Hardman and Aitkenhead equation [1.14 × (Paco2- Etco2)/Paco2 - 0.005].
intrapulmonary shunt | 20 minutes after iloprost inhalation (T2)
  -Shunt fraction (Qs/Qt) was calculated using the following formula: Qs/Qt = (CcO2-CaO2)/(CcO2-CvO2), (1)
  -whereby:
  * CaO2 = (PaO2 x 0.0031) + (Hemoglobin x 1.36 x SaO2), (2)
  * CvO2 = (PvO2 x 0.0031) + (Hemoglobin x 1.36 x SvO2), (3)
  * CcO2 = ([FiO2 x (PB - PH2O) - PaCO2/Respiratory quotient] x 0.0031) + (Hemoglobin x 1.36), (4)
  * PB is the barometric pressure (760 mmHg), the PH2O is 47 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No